CLINICAL TRIAL: NCT01121471
Title: Supplementation With Conjugated Linoleic Acid (CLA) as Complementary Therapy in the Management of Type 2 Diabetes Mellitus (Women's Diabetes Study)
Acronym: WDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Cognis (Industry)
Responsible Party: Martha A. Belury, The Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003H0122
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; conjugated linoleic acid
MeSH Terms: conditions — Diabetes Mellitus | interventions — Linoleic Acids, Conjugated; Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Safflower Oil (Placebo Comparator): 8.0 g/day safflower oil
  Interventions: Dietary Supplement: Safflower OIl
- CLA 6.4g/day (Experimental): Conjugated linoleic acid at a dose of 6.4g/day in a supplement with a total of 8.0g oil
  Interventions: Dietary Supplement: Conjugated Linoleic Acid (CLA)

INTERVENTIONS:
Dietary Supplement: Conjugated Linoleic Acid (CLA) — 6.4 g CLA/day, capsule form, for 16 week arms
  Arms: CLA 6.4g/day
Dietary Supplement: Safflower OIl — 8.0g/day safflower oil
  Arms: Safflower Oil

SUMMARY:
The purpose of this study is to determine the role of CLA as a complementary therapy to improve body composition, glucose tolerance, fasting plasma glucose and insulin, and hemoglobinA1c (HbA1c) in subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
The design is a double-blind, placebo-controlled, crossover study conducted at a single site. The primary variable is a change from baseline to Week 16 in plasma glucose area under the curve during a three-hour oral glucose tolerance test. Secondary variables include changes in fasting levels of glucose and insulin, glucose tolerance, hemoglobinA1c, hepatic enzymes, adipocytokines, blood lipid profile, and body composition. Supporting endpoints include dietary intake, physical activity, fatty acids, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Type 2 diabetes mellitus
* obese
* postmenopausal
* HbA1c >6.49 and <14.1

Exclusion Criteria:

* use of tobacco
* substance abuse
* impaired cognitive function
* renal disease
* abnormal liver function
* gastrointestinal diseases
* use of exogenous insulin
* use of hormone replacement therapy currently or within past 6 months
* pacemaker/defibrillator

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-12; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
change in plasma glucose AUC | baseline and week 16
  significant change in plasma glucose AUC (0-3 h) from baseline to Week 16.

SECONDARY OUTCOMES:
change in insulin sensitivity | baseline and every 4 weeks until week 16
change in glucose tolerance | baseline and every 4 weeks for 16 weeks
change in HbA1c | baseline and week 16
change in blood lipid profile | baseline and every 4 weeks for 16 weeks
change in serum adipocytokines | baseline and every 4 weeks for 16 weeks
change in hepatic enzymes | baseline and every 4 weeks for 16 weeks
change in body composition | baseline and every 4 weeks for 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martha A. Belury, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Norris LE, Collene AL, Asp ML, Hsu JC, Liu LF, Richardson JR, Li D, Bell D, Osei K, Jackson RD, Belury MA. Comparison of dietary conjugated linoleic acid with safflower oil on body composition in obese postmenopausal women with type 2 diabetes mellitus. Am J Clin Nutr. 2009 Sep;90(3):468-76. doi: 10.3945/ajcn.2008.27371. Epub 2009 Jun 17. PMID 19535429